CLINICAL TRIAL: NCT00550641
Title: Pool-based Exercise in Fibromyalgia Management: a Prospective Randomized Comparison Between Stretching and Ai Chi
Brief Title: Pool-based Exercise in Fibromyalgia Management
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad de Granada (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML-2006
Record Dates: First submitted 2007-10-26; First posted 2007-10-30 (Estimated); Last update posted 2010-04-06 (Estimated); Status verified 2007-09

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia; pool-based exercise
MeSH Terms: conditions — Fibromyalgia | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Other: physical therapy
- 2 (Experimental)
  Interventions: Other: physical therapy

INTERVENTIONS:
Other: physical therapy — physical therapy in warm pool performing stretching
  Arms: 1
Other: physical therapy — physical therapy in warm pool performing Ai Chi
  Arms: 2

SUMMARY:
Pharmacologic treatment remains the primary therapeutic approach in fibromyalgia management, but different non-pharmacologic measures, especially physical therapies and psychologically-based interventions, have also shown to be effective in the treatment of this disease. The objective of the present randomized controlled trial is to compare the efficacy and tolerability of two different modalities of active low-impact exercise in warm water: stretching and Ai Chi. Each group of patients will receive 18 physiotherapy sessions lasting 60 minutes and will be evaluated at baseline, at treatment termination, and after 4 and 12 weeks of follow up. Main outcome measures are the Fibromyalgia Impact Questionnaire (FIQ) and the Pittsburgh Sleep Quality Index (PSQI). Secondary outcome measures include the Beck Depression Inventory (BDI), the State and Trait Anxiety Inventory (STAI), and the SF-12 Health Survey (SF-12. Data analysis will be done using repeated measures ANOVA, unpaired Student's t test, and effect sizes' estimation (ES).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of fibromyalgia according to the ACR criteria
* 18 years or older
* written informed consent to participate

Exclusion Criteria:

* unable to tolerate warm chlorinated water
* associated medical condition contraindicating exercise in warm water

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2006-03; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Improvement in fibromyalgia symptomatology | 18 weeks

SECONDARY OUTCOMES:
Improvement in sleep, depressive and anxiety symptomatology and quality of life | 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Elena P. Calandre, Study Director — Professor of Clinical Pharmacology; Mª Luz Rodriguez-Claro, Principal Investigator — physiotherapist
Locations (1):
- Hospital Universitario "Virgen de las Nieves", Granada, Granada, Spain

REFERENCES:
- [Result] Calandre EP, Rodriguez-Claro ML, Rico-Villademoros F, Vilchez JS, Hidalgo J, Delgado-Rodriguez A. Effects of pool-based exercise in fibromyalgia symptomatology and sleep quality: a prospective randomised comparison between stretching and Ai Chi. Clin Exp Rheumatol. 2009 Sep-Oct;27(5 Suppl 56):S21-8. PMID 20074435